CLINICAL TRIAL: NCT03141515
Title: Sonographic Assessment of Postural Lung Recruitment in Pediatric Patients Under General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Privado de Comunidad de Mar del Plata (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HospitalPC
Record Dates: First submitted 2017-04-17; First posted 2017-05-05 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2017-05

CONDITIONS: Collapsed Lung
Keywords: lung ultrasound; recruitment maneuver; atelectasis; children
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): After anesthesia induction patients received lung recruitment maneuver using pressure-control ventilation with a patient in supine position with 10 cmH2O level of positive end-expiratory pressure PEEP during 180 seconds. Lung ultrasound examination will be performed at two different times-point immediately after induction and after recruitment maneuver to monitor lung aeration.
  Interventions: Device: Lung ultrasound
- Recruitment maneuver group (Experimental): Patients received lung recruitment maneuver with postural changes of lateral decubitus using pressure-control ventilation, 10 cmH2O level of PEEP in left and in right lateral decubitus during 90 seconds in each one. Lung ultrasound examination will be performed at two different times-point immediately after induction and after recruitment maneuver to monitor lung aeration.
  Interventions: Device: Lung ultrasound

INTERVENTIONS:
Device: Lung ultrasound — Lung ultrasound examination at two different times-point immediately after induction and after recruitment maneuver to monitor lung aeration.

SUMMARY:
Anesthesia-induced atelectasis is a well-known entity observed in approximately 68-100% of pediatric patients undergoing general anesthesia. The collapse of dependent lung zones starts with anesthesia induction but can persist for hours or even days after surgery.

Lung collapse is a pressure-dependent phenomenon. Each acinus has a critical closing pressure, i.e., the minimum transpulmonary pressure (Ptp) below that the acinus begins to collapse. While airway pressure is homogeneously distributed within all lung units, Pleural pressure increases along the vertical gravitational vector because of the lung's weight. As a consequence, the decreased Ptp in the dependent zones promotes collapse. This means that patients in the supine position suffer from increasing closing pressures in the ventral to dorsal direction.

Alveolar recruitment maneuvers recruit collapsed alveoli, increase gas exchange, and improve arterial oxygenation.

The investigators hypothesized that in children with anesthesia-induced atelectasis, postural changes have recruiting effects and improve lung aeration assessed by lung ultrasound.

DETAILED DESCRIPTION:
Compare lung aeration between two different lung recruitment strategies (recruitment maneuvers in supine position and recruitment maneuvers with postural changes of lateral decubitus with 10 cmH2O level of positive-end expiratory pressure (PEEP) during 180 seconds; in pediatric patients scheduled for surgery under general anesthesia using ultrasound imaging and a four-point-aeration score to assess the lung aeration.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent by parents.
* Patients aged 6 months to 5 years old
* Scheduled for surgery under general anesthesia with tracheal intubation with atelectasis assessed by lung ultrasound after anesthesia induction.
* American Society of Anesthesiologists classification: physical status I-II

Exclusion Criteria:

* Acute airway infection
* Cardiovascular or pulmonary disease
* Previous thoracic procedure

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-01-05 (Actual); Study Completion 2018-01-05 (Actual)

PRIMARY OUTCOMES:
Lung aeration | Intraoperative
  Compare lung aeration between two different lung recruitment strategies (recruitment maneuvers in supine position with 10 cmH2O level of PEEP during 180 seconds and recruitment maneuvers with postural changes of lateral decubitus: 10 cmH2O level of PEEP in left and in right lateral decubitus during 90 seconds in each one) in pediatric patients scheduled for surgery under general anesthesia using ultrasound imaging and a four-point-aeration score to assess the lung aeration (0 = normal lung, 1 = moderate aeration loss, 2 = severe aeration loss, 3 = complete aeration loss and consolidation).

SECONDARY OUTCOMES:
Peripheral arterial oxygenation by pulse oximetry (SPO2%) | Intraoperative
  The SPO2 % will be recorded before and after recruitment manoeuvre.
Respiratory mechanics | Intraoperative
  Intra-operative ventilator data will be recorded to measure respiratory mechanics such as dynamic and statistic compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia M Acosta, MD, Principal Investigator — Hospital Privado de Comunidad
Locations (1):
- Cecilia M. Acosta, Mar del Plata, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No